CLINICAL TRIAL: NCT02002988
Title: Endomyocardial Botulinum Toxin Injection Can Prevent Drug-Resistant Paroxysmal Atrial Fibrillation: Pilot Study
Brief Title: Botulinum Toxin Injection Prevent Paroxysmal Atrial Fibrillation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT_PAF01
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BT injection (Experimental)
  Interventions: Procedure: endomyocardial BT injection

INTERVENTIONS:
Procedure: endomyocardial BT injection

SUMMARY:
The aim of this prospective non-randomized study was to assess the efficacy and safety of endomyocardial botulinum toxin injection in projections of main ganglionated plexuses of left atrium for preventing drug-resistant paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* drug-resistant PAF

Exclusion Criteria:

* Previous heart surgery and AF ablation procedure
* Emergency CABG
* Unstable angina or heart failure
* Persistent AF, AF at the time of screening (planned Maze procedure or pulmonary vein isolation)
* Use of I or III antiarrhythmic drugs within 5 elimination half-lives of the drug (or within 2 months for amiodarone)
* Requiring concomitant valve surgery
* Left ventricle ejection fraction <35%
* Left atrial diameter >55 mm
* Unwillingness to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
serious adverse events | 1 year

SECONDARY OUTCOMES:
number of paroxysms | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru